CLINICAL TRIAL: NCT03339804
Title: Neurovascular Changes Provoked by Acute Administration Doxorubicin and Cyclophosphamide in Patients With Breast Cancer
Brief Title: Neurovascular Changes Induced by Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SDC 4227/15/054
Record Dates: First submitted 2017-10-25; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer; Chemotherapeutic Toxicity
Keywords: Chemotherapy; Muscle sympathetic nervous activity; Blood flow; Endothelial microparticles
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy (Experimental): Infusion of doxorubicin and cyclophosphamide
  Interventions: Other: Chemotherapy

INTERVENTIONS:
Other: Chemotherapy — In chemoteraphy session, doxorubicin (60 mg/m2) and cyclophosphamide (600mg/m2) were administred in 45 min
  Other Names: Doxorubicin and cyclophosphamide

SUMMARY:
The purpose of the present study was to test the hypothesis that doxorubicin and cyclophosphamide adjuvant chemotherapy (CHT) acutely induces neurovascular and hemodynamic changes in patients with breast cancer. To test this hypothesis, women with breast cancer (stage II-III) underwent two experimental sessions, saline (SL) and CHT. In the CHT session, doxorubicin (60 mg/m2) and cyclophosphamide (600mg/m2) were administred in 45 min. In the SL session, a matching saline volume to that of the CHT session was infused over 45 min.

DETAILED DESCRIPTION:
The purpose of the present study was to test the hypothesis that doxorubicin and cyclophosphamide adjuvant chemotherapy (CHT) acutely induces neurovascular and hemodynamic changes in patients with breast cancer. To test this hypothesis, the patients were submitted in two experimental sessions, saline and chemotherapy, respectively. Saline Session. After fasting for 2 hours and abstaining from caffeine for 24 hours, the patients were positioned in a supine position. An intra-venous catheter was placed into the brachial venous in the contralateral arm of the breast surgery. Microelectrodes were positioned for MSNA measures in right leg, cuffs were placed around the leg for blood flow assessments and finger cuff was placed in 3 finger of hand for measurement of hemodynamic variables. After the instrumentation, an interval of 10 minutes was allowed, followed by blood sample collections for measurement of MPEs and, hemodynamic and neurovascular measures by period of 15 minutes (pre-infusion). Then, dexamethasone 20 mg and ondansetron 8 mg were administered i.v., followed by saline 0,09%, during 45 minutes. During saline infusion were continuously measured the neurovascular and hemodynamic variables. Finally, after saline administration, another blood sample was collected for MPEs dosing, followed by continuous measurement of hemodynamic and neurovacular variables by 15 minutes period (Figure 1).

Chemotherapy session. After a 2 to 3 day-interval, the patients were again positioned in a supine position in a temperature-controlled room (22oC). An intra-venous catheter was placed into the brachial venous in the contralateral arm of the breast surgery. Then, microelectrodes were positioned in the contralateral leg of the first session for MSNA measures. Likewise, cuffs were placed around the contralateral leg of the first protocol for blood flow assessments. After the instrumentation, an interval of 10 minutes was allowed, followed by blood sample collections and basal hemodynamic and neurovascular measures. Then, dexamethasone 20 mg and ondansetron 8 mg were administered, i.v., followed by doxorubicin and cyclophosphamide, during 45 minutes. During doxorubicin and cyclophosphamide infusions were continuously measured the neurovascular and hemodynamic variables. Finally, after doxorubicin plus cyclophosphamide administration, another blood sample was collected for EMPs dosing, followed by continuous measurement of hemodynamic and neurovacular variables by 15 minutes period

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients and prescription of adjuvant chemotherapy with antracycline and cyclophosphamide

Exclusion Criteria:

* Metastic disease
* Hypercholesterolemia
* Diabetes
* Hypertension
* Severe lymphedema
* Renal insufficient
* Heart failure
* Chronic liver disease
* Obesity, and treatment with some medications that inhibit cardiotoxicity, as beta-blocker angiotensin converting enzyme, statin, losartan and antioxidants.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Neural change induced by chemoterapy | 10 min
  Increase of muscle nerve sympathetic activivity

SECONDARY OUTCOMES:
Vascular change induced by chemoterapy | 10 min
  Decrease of blood flow

OTHER OUTCOMES:
Hemodynamic change induced by chemoterapy | 10 min
  Increase of blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Negrão, Principal Investigator — University of Sao Paulo
Locations (1):
- Heart Institute, São Paulo, Cerqueira Cesar, Brazil

IPD SHARING:
Plan to Share IPD: No